CLINICAL TRIAL: NCT02674802
Title: Reinfection After Eradication of Helicobacter Pylori Infection in Adult :A National Multicentre Study
Brief Title: Reinfection After Eradication of Helicobacter Pylori Infection
Acronym: RAEHPI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Nanchang University (Other)
Responsible Party: Principal Investigator, Lingyu Luo, Physician-in-charge, The First Affiliated Hospital of Nanchang University
Other Study IDs: Affiliated Hospital of NCU
Record Dates: First submitted 2016-02-02; First posted 2016-02-04 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-02

CONDITIONS: Bacterial Infection Due to Helicobacter Pylori (H. Pylori); Eradication Therapy of Helicobacter Pylori; Detection of Helicobacter Pylori
Keywords: Reinfection; Eradication therapy; C-urea breath test; Helicobacter Pylori
MeSH Terms: conditions — Reinfection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Retrospective study: People who has successfully eradicated helicobacter pylori more than six months detected helicobacter pylori by the C-urea breath test in order to evaluate the reinfection.
- Prospective study: People who has infected helicobacter pylori received regular eradication therapy after the 4 weeks, 8 weeks and 6 months detected helicobacter pylori by the C-urea breath test in order to prospect the reinfection .

SUMMARY:
Helicobacter pylori is closely related with gastritis, peptic ulcer, gastric cancer and gastric MALT lymphoma, and it may participate in a variety of parenteral diseases. Infection rates of Helicobacter pylori is still high, so effectively eradication is necessary. At present, the eradication therapy has achieved very good curative effect. However, relapse after eradication is unoptimistic. This study has made an analysis for reinfection after eradication of Helicobacter pylori Infection include the retrospective and prospective studies, aims to explore the epidemiological data and related risk factors of Hp reinfection in China.

DETAILED DESCRIPTION:
In the retrospective study,we choose the people received regular eradication therapy, successfully eradicated helicobacter pylori more than six months, but 4 to 8 weeks after drug withdrawal ,the detection result of helicobacter pylori were negative to ensure that the results of the study is the reinfection, not residual. Even more noteworthy is during the treatment and detection again, the patients must not received any eradication therapy of Hp. What's more , before the detection, they also has not used antibiotics, bismuth agent and the traditional Chinese medicine with antibacterial effect in 1 monthor and has not used H2RA and PPI in 2 weeks to prevent affecting the accuracy of the results. At the same time, we also investigated the patient's general situation, conomic conditions, living conditions, personal health and lifestyle to explore related risk factors of Hp reinfection in China. In the prospective study, we detected Hp by C-UBT after regular eradication therapy of Hp for 4 weeks, 8 weeks and 6 months to prospect the reinfection of Hp.It also can make up the defects of retrospective study.

ELIGIBILITY:
Inclusion Criteria:

-1、Retrospective study：

1. Received regular eradication therapy, 4 to 8 weeks after drug withdrawal , detected of helicobacter pylori and the results were negative
2. Eradication program and original disease is unlimited
3. Without any eradication therapyof Hp during the treatment and detection again
4. before the detection has not used antibiotics, bismuth agent and the traditional Chinese medicine with antibacterial effect in 1 monthor and has not used H2RA and PPI in 2 weeks.

2、Prospective study

1. Infected with H. pylori that detected by C-UBT
2. With out alimentary tract hemorrhage,ulceration and complications of eradication
3. Eradication program and original disease is unlimited

Exclusion Criteria:

1. Pregnancy or breast-feeding women
2. With the major disease which would influence the research such as liver disease, heart disease, kidney disease, malignant tumor and alcohol poisoning
3. Participated in other drug research in the past three months
4. The patient can't express himself correctly such as mental illness and severe neurosis and can't cooperation this test

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In the retrospective study,people who has infected helicobacter pylori and successfully eradicated it more than six months detected helicobacter pylori by the C-urea breath test in order to evaluate the reinfection In the prospective study,people who has infected helicobacter pylori received regular eradication therapy after the 4 weeks, 8 weeks and 6 months detected helicobacter pylori by the C-urea breath test in order to prospect the reinfection
Sampling Method: Non-Probability Sample
Enrollment: 3500 (Estimated)
Dates: Start 2015-12; Primary Completion 2016-03 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Helicobacter Pylori Infection | six months
  Retrospective study
Helicobacter Pylori Infection | After regular eradication therapy of Hp for 4 weeks, 8 weeks and 6 months
  Prospective study

CONTACTS AND LOCATIONS:
Overall Officials: Nonghua Lv, MD, Study Chair — The First Affiliated Hospital of Nanchang University
Locations (1):
- Affiliated Hospital of Nanchang University, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Malfertheiner P, Megraud F, O'Morain CA, Atherton J, Axon AT, Bazzoli F, Gensini GF, Gisbert JP, Graham DY, Rokkas T, El-Omar EM, Kuipers EJ; European Helicobacter Study Group. Management of Helicobacter pylori infection--the Maastricht IV/ Florence Consensus Report. Gut. 2012 May;61(5):646-64. doi: 10.1136/gutjnl-2012-302084. PMID 22491499
- [Background] Silva FM, Navarro-Rodriguez T, Barbuti RC, Mattar R, Hashimoto CL, Eisig JN. Helicobacter pylori reinfection in Brazilian patients with peptic ulcer disease: a 5-year follow-up. Helicobacter. 2010 Feb;15(1):46-52. doi: 10.1111/j.1523-5378.2009.00734.x. PMID 20302589
- [Background] Benajah DA, Lahbabi M, Alaoui S, El Rhazi K, El Abkari M, Nejjari C, Amarti A, Bennani B, Mahmoud M, Ibrahimi SA. Prevalence of Helicobacter pylori and its recurrence after successful eradication in a developing nation (Morocco). Clin Res Hepatol Gastroenterol. 2013 Nov;37(5):519-26. doi: 10.1016/j.clinre.2013.02.003. Epub 2013 Apr 6. PMID 23567104
- [Background] Take S, Mizuno M, Ishiki K, Imada T, Okuno T, Yoshida T, Yokota K, Oguma K, Kita M, Okada H, Yamamoto K. Reinfection rate of Helicobacter pylori after eradication treatment: a long-term prospective study in Japan. J Gastroenterol. 2012 Jun;47(6):641-6. doi: 10.1007/s00535-012-0536-9. Epub 2012 Feb 17. PMID 22350696
- [Background] Archimandritis A, Balatsos V, Delis V, Manika Z, Skandalis N. "Reappearance" of Helicobacter pylori after eradication: implications on duodenal ulcer recurrence: a prospective 6 year study. J Clin Gastroenterol. 1999 Jun;28(4):345-7. doi: 10.1097/00004836-199906000-00012. PMID 10372933
- See also: the First Affiliated Hospital of Nanchang University — http://www.cdyfy.com/